CLINICAL TRIAL: NCT00302601
Title: The Acute Pulmonary Embolism 1 (APE 1) Trial: Prospective Investigation of Scintigraphic Diagnosis and Pathophysiology of Right Heart Strain
Brief Title: Study of Diagnosis and Pathophysiology of Pulmonary Embolism (APE 1 Trial)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics failure and staff/scanner shortage
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Søren Hess, MD, Chief physician, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 70
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Embolism; Right Heart Strain
Keywords: Pulmonary embolism; Right heart strain; Lung scintigraphy; Pulmonary angiography
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- None relevant (Other): Not relevant
  Interventions: Procedure: Scintigraphic interpretation

INTERVENTIONS:
Procedure: Scintigraphic interpretation — Not relevant

SUMMARY:
The purpose of this study is to

* investigate which method and criterion for diagnosing pulmonary embolism is the best and
* determine the relationship between blood vessel constriction and clot size in patients developing heart failure

DETAILED DESCRIPTION:
INTRODUCTION This project assesses both scintigraphic diagnosis and the pathophysiology of right heart strain in acute pulmonary embolism. The primary purposes are to validate various scintigraphic methods with pulmonary angiography as the standard of reference (purpose A). Furthermore, this project examines the relative contributions of 1) vascular obstruction, 2) vasoactive mediators, and 3) co-morbidity to the generation of right heart strain (purpose B).

BACKGROUND FOR PURPOSE A Acute pulmonary embolism is a life threatening condition. Early intervention can be lifesaving but treatment is associated with severe side effects. Thus, establishing accurate diagnosis is necessary. Clinical presentation and physical examination have proven insufficient for this purpose. This is also true for basic diagnostic investigations, e.g. electrocardiography, arterial blood gas analysis and chest x-ray, which are considered standard tests in patients with symptoms consistent with cardiopulmonary disease.

For several decades lung scintigraphy has been considered a cornerstone in the diagnosis of acute pulmonary embolism. Planar two-dimensional images of the pulmonary perfusion are obtained using a gamma camera after intravenous injection of radiolabelled microparticles, depicting perfusion defects caused by e.g. a pulmonary embolus. Similarly, ventilatory function can be assessed two-dimensionally by planar scintigraphic imaging following inhalation of a radioactive gas or aerosol. Lung scintigraphy has certain limitations, primarily related to image interpretation. The PIOPED criteria, based on the combined ventilation-perfusion scintigraphy, have gained global acceptance, but are often inconclusive and give rise to misunderstandings. A different set of interpretation criteria, provided by the PISA-PED study group, are based solely on perfusion imaging. Opposite the PIOPED criteria, PISA-PED criteria are always conclusive and exhibits both high sensitivity and specificity. The latter have, however, not gained the same widespread acceptance as the PIOPED criteria. It remains uncertain which set of criteria is the better to confirm or exclude the diagnosis of acute pulmonary. A prospective trial evaluating both PIOPED criteria (original and revised) and PISA-PED criteria against a valid standard of reference therefore seems appropriate.

The more resource demanding single photon emission computed tomography (SPECT) has recently been subject to renewed interest in the diagnosis of acute pulmonary embolism, but it remains unclear whether this technique offers additional information compared to conventional planar imaging. SPECT offers three-dimensional images, but otherwise the technique is similar to the methods described for planar images. Combining the PISA-PED criteria and SPECT imaging has not yet been tested in a prospective trial, but it seems highly relevant.

Since the diagnosis is often suspected several times in the same patient, the ability to distinguish acute and chronic changes in the scintigrams are essential. It is, however, unclear to what extend and how fast the scintigraphic changes resolve. This has great implications in scintigraphic control of patients recovering from acute pulmonary embolism.

A trial regarding the statements above requires a reliable method to test whether the patient is suffering from acute pulmonary embolism or not: a standard of reference. Pulmonary angiography is traditionally conceived as the standard of reference in acute pulmonary embolism, but only a few newer studies employ this technique.

BACKGROUND FOR PURPOSE B Right heart strain is a common finding in acute pulmonary embolism. It is a result of the sudden increase in pressure in the pulmonary circulation. Ultrasonographic examination of the heart by echocardiography is suitable to demonstrate this condition and this finding in a patient with acute pulmonary embolism is associated with a considerably worse prognosis. The degree of right heart strain is not exclusively determined by extension or size of the embolus. There is substantial evidence of the influence of both co-morbidity and the release of vasoactive mediators on the extend of right heart strain. The exact interplay between these three factors is not completely understood in humans. Albeit, this can have significant implications on therapy, since pharmacological manipulation of vascular tone in the pulmonary circulation is possible. This treatment is, however, not without risk, and no well-designed study has yet addressed these issues in patients with acute pulmonary embolism. Several case reports on successful treatment with vasodilation, e.g. with inhaled nitric oxide, have been published. A more profound understanding of the etiology of acute right heart failure in acute pulmonary embolism is therefore desirable. What is the individual contribution of 1) clot burden, 2) release of vasoactive mediators, and 3) co-morbidity?

Recently, acute pulmonary embolism has been divided into three categories depending on clinical presentation and echocardiographic findings: 1) massive; in which the patient suffers from cardiac arrest or cardiogenic shock. Most authorities agree that these patients should be treated with fibrinolytic agents. 2) Non-massive; with no signs of shock or right heart strain. In these patients there is no indication for fibrinolytic agents. 3) Sub-massive; with no manifestations of shock but echocardiographic findings consistent with right heart strain. The indication for fibrinolytic treatment in this last group is unresolved. This study will address whether simple methods, e.g. peripheral blood sampling and perfusion scintigraphy can determine the primary mechanism in the generation of right heart strain in the individual patient.

A later (not yet planned) intervention study based on the abovementioned knowledge could then address the following question: Should the patient with sub-massive pulmonary embolism receive treatment with fibrinolytic agents (in the case of major clot burden and minor degree of pulmonary vasoconstriction) or vasodilators (minor clot burden, major degree of pulmonary vasoconstriction)?

ELIGIBILITY:
Inclusion Criteria:

* Referred from clinical departments at Odense University Hospital
* Referred to the Departments of Nuclear Medicine or Radiology for diagnostic evaluation of suspected pulmonary embolism
* Referred for lung scintigraphy, spiral computer tomography, or pulmonary angiography

Exclusion Criteria:

* Age below 18
* Contrast allergy
* Pregnancy
* S-Creatinine above 200 micromol/L
* Metformin treatment
* Fibrinolytic or surgical therapy between examinations
* No informed consent
* Withdrawn consent
* Failed logistics (more than 24 hours between examinations)
* No conclusive pulmonary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Purpose A: Specificity, sensitivity, predictive values, and observer variation for scintigraphic procedures | 2006-2012
Purpose B: Blood concentrations of vasoactive substances, clot size on scintigram. | 2006-2012

CONTACTS AND LOCATIONS:
Overall Officials: Poul Henning Madsen, MD, Principal Investigator — Department of Nuclear Medicine, Odense University Hospital; Soeren Hess, MD, Principal Investigator — Department of Nuclear Medicine, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No